CLINICAL TRIAL: NCT06926751
Title: A Multicenter, Randomized, Controlled Study of Telpegfilgrastim Versus Filgrastim for Secondary Prevention of Chemotherapy-Induced Neutropenia in Children and Adolescents With Solid Tumors Receiving High-Intensity Chemotherapy Regimens
Brief Title: Telpegfilgrastim vs Filgrastim for Secondary Prevention of Chemotherapy-Induced Neutropenia in Pediatric Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, SIDAN LI, Prof, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PJ-B-241113
Record Dates: First submitted 2025-04-06; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumors; Children; Adolescent; Chemotherapy Induced Neutropenia
MeSH Terms: interventions — Filgrastim; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, open-label, randomized controlled trial. It plans to enroll 132 children and adolescent patients with malignant solid tumors receiving high-density chemotherapy regimens. Patients will be randomized in a 3:1 ratio to receive Telpegfilgrastim or filgrastim for the prevention of chemotherapy-induced neutropenia (CIN), with observation of efficacy and safety in both groups. Patient data from all centers will be collected through an Electronic Data Capture (EDC) system.
  The trial employs a stratified randomization method based on subjects' age (6-12 years, 13-18 years, and 19-24 years). After signing the informed consent form, each subject will be assigned a unique screening number for identification throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telpegfilgrastim (Experimental): Receive subcutaneous injections of Telpegfilgrastim (33 μg/kg, single dose) 24 hours after each chemotherapy cycle
  Interventions: Drug: Telpegfilgrastim Injection
- Filgrastim (Active Comparator): Receive subcutaneous injections of Filgrastim (5 μg/kg/day, multiple doses) 24 hours after each chemotherapy cycle
  Interventions: Drug: filgrastim

INTERVENTIONS:
Drug: Telpegfilgrastim Injection — subcutaneous injections of Telpegfilgrastim (33 μg/kg, single dose) 24 hours after each chemotherapy cycle
  Other Names: Y-branched pegylated recombinant human granulocyte colony stimulating factor; YPEG-G-CSF; Peijin
  Arms: Telpegfilgrastim
Drug: filgrastim — subcutaneous injections of Filgrastim (5 μg/kg/day, multiple doses) 24 hours after each chemotherapy cycle
  Other Names: Recombinant Human Granulocyte-Colony Stimulating Factor; rhG-CSF; Topneuter
  Arms: Filgrastim

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Telpegfilgrastim (a PEGylated recombinant human granulocyte colony-stimulating factor, PEG-rhG-CSF) compared to Filgrastim (short-acting rhG-CSF) in preventing chemotherapy-induced neutropenia (CIN) in children and adolescents aged 6-24 years with malignant solid tumors receiving high-intensity chemotherapy regimens. The main questions it aims to answer are:

* Does Tuopefilgrastim reduce the incidence of febrile neutropenia (FN) in the first chemotherapy cycle (Cx+1) compared to Filgrastim?
* How do the two treatments compare in terms of duration and severity of neutropenia, chemotherapy delays/dose reductions, antibiotic use, and bone pain incidence? Researchers will compare the Telpegfilgrastim group (3:1 ratio, 99 participants) with the Filgrastim group (33 participants) to determine if Telpegfilgrastim demonstrates superior efficacy and safety.

Participants will:

* Receive subcutaneous injections of either Telpegfilgrastim (33 μg/kg, single dose) or Filgrastim (5 μg/kg/day, multiple doses) 24 hours after each chemotherapy cycle.
* Undergo blood tests, physical exams, and temperature monitoring during follow-up visits.
* Be assessed for bone pain severity using age-appropriate scales (FLACC or Wong-Baker).
* Complete two chemotherapy cycles with close safety and efficacy monitoring.

DETAILED DESCRIPTION:
This multicenter, randomized, open-label, controlled clinical trial evaluates the efficacy and safety of Telpegfilgrastim, a novel 40kD Y-branched PEGylated recombinant human granulocyte colony-stimulating factor (PEG-rhG-CSF), compared to Filgrastim (short-acting rhG-CSF) in preventing chemotherapy-induced neutropenia (CIN) among pediatric and adolescent patients (aged 6-24 years) with malignant solid tumors receiving high-intensity chemotherapy. The study employs a two-phase adaptive design: Phase 1 involves 20 participants (15 in the Telpegfilgrastim arm, 5 in the Filgrastim arm) to assess preliminary pharmacokinetics (PK) and safety, including drug half-life (71.7 ± 23 hours for Telpegfilgrastim vs. 3.5-4 hours for Filgrastim) and neutrophil recovery dynamics, with potential dose adjustments before progressing to Phase 2. The full trial enrolls 132 participants randomized 3:1 (99 vs. 33), stratified by age subgroups (6-12, 13-18, 19-24 years) to account for developmental variations in drug metabolism. Telpegfilgrastim is administered as a single subcutaneous injection (33 μg/kg, max 2 mg) 24 hours post-chemotherapy, leveraging its prolonged activity from Y-shaped PEGylation, while Filgrastim requires daily injections (5 μg/kg/day) until absolute neutrophil count (ANC) recovers to ≥10.0×10⁹/L. Concomitant use of other myelostimulatory agents (e.g., GM-CSF, trilaciclib) is prohibited to isolate treatment effects.

Neutrophil monitoring includes ANC measurements at baseline and days 7, 9, 11, 13, 15, and 21 (±1 day) post-chemotherapy using standardized hematology analyzers. Febrile neutropenia (FN) is strictly defined as ANC <0.5×10⁹/L (Grade 4) or ANC 0.5-<1.0×10⁹/L (Grade 3) with anticipated decline to <0.5×10⁹/L within 48 hours, accompanied by axillary temperature ≥37.7°C sustained for ≥1 hour. Bone pain, a key safety focus, is assessed using age-specific tools: the FLACC scale (Face, Legs, Activity, Cry, Consolability; 0-10) for children <8 years and the Wong-Baker Faces Pain Rating Scale (0-10) for older participants. Exploratory analyses evaluate bone metabolism through serial serum osteocalcin (osteoblast activity marker) and RANKL/OPG ratio (osteoclast regulation) measurements at baseline, day 7, and day 21, with optional bone marrow aspirates to assess hematopoietic stem/progenitor cell (HSPC) mobilization efficiency.

Data management utilizes a validated electronic data capture (EDC) system with real-time entry and automated queries for anomalies, complemented by source data verification (SDV) for ≥20% of cases, prioritizing primary endpoints and serious adverse events (SAEs). Sample size (132 participants) is calculated based on prior pediatric FN incidence rates (45% PEG-rhG-CSF vs. 75% rhG-CSF), with α=0.05, 80% power, and 20% attrition. Statistical analyses employ the Full Analysis Set (FAS, intent-to-treat) and Per-Protocol Set (PPS), using ANOVA or nonparametric tests for continuous variables (e.g., ANC recovery time) and Chi-square/Fisher's exact tests for categorical outcomes (e.g., FN incidence), adjusted for age, tumor type, and chemotherapy regimen. Safety analyses include all participants receiving ≥1 dose (Safety Set), with SAEs reported per ICH-GCP and China NMPA guidelines, monitored by an independent Data Safety Monitoring Board (DSMB).

Ethical compliance is ensured through institutional review board (IRB) approvals at all 16 participating centers, emphasizing informed consent/assent for adolescents, anonymized biological sample storage (≤5 years post-trial), and voluntary withdrawal rights. The trial's innovation lies in its focus on pediatric PK/PD profiling, addressing faster drug clearance in children, and evaluating long-term skeletal safety via bone metabolism biomarkers-critical for growing populations. By comparing next-generation PEG-rhG-CSF with conventional rhG-CSF, this study aims to refine global supportive care guidelines for pediatric oncology, balancing efficacy and safety in high-intensity chemotherapy settings.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed malignant solid tumor requiring high-intensity chemotherapy, with ≥2 remaining chemotherapy cycles, and either:

   * Previous febrile neutropenia(FN) or dose-limiting neutropenia in the prior chemotherapy cycle without prophylactic granulocyte colony-stimulating factor (G-CSF);
   * Previous FN or dose-limiting neutropenia in the prior chemotherapy cycle despite prophylactic G-CSF.
2. Age ≥6 to ≤24 years.
3. Eastern Cooperative Oncology Group Performance Status ≤1.
4. Normal bone marrow hematopoietic function: hemoglobin ≥75 g/L, white blood cell count ≥3.0×10^9/L, platelets ≥80×10^9/L, and neutrophils ≥1.5×10^9/L.
5. Anticipated survival ≥8 months.
6. Willing to participate, with written informed consent signed by the patient or legal guardian.

Exclusion Criteria:

1. Bone marrow involvement at screening.
2. Uncontrolled localized or systemic infection.
3. Known hypersensitivity to Telpegfilgrastim, recombinant human granulocyte-colony stimulating factor(rhG-CSF), or other pegylated recombinant human granulocyte colony stimulating factor(PEG-rhG-CSF) agents.
4. Concurrent participation in any other investigational drug or device trial.
5. Severe organ dysfunction: total bilirubin, alanine aminotransferase(ALT), or aspartate transaminase(AST) >2.5 × upper limit of normal(ULN) (or >5 × ULN in patients with liver metastases), serum creatinine >5 × ULN.
6. Severe psychiatric disorders affecting informed consent provision or adverse event assessment.
7. Any condition deemed by the investigator to compromise patient safety or interfere with study outcomes, including risks from the investigational product or confounding adverse event evaluation.

Ages: 6 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of febrile neutropenia in Cycle 1 | 21-28 days
  Incidence of febrile neutropenia in Cycle 1 (i.e., the first chemotherapy cycle post-enrollment)

SECONDARY OUTCOMES:
Incidence of grade 3 neutropenia during Cycles 1-2 | 42-56 days
  Incidence of grade 3 neutropenia (absolute neutrophil count<1.0×10^9/L) during Cycles 1-2
Time to recovery of grade 3 neutropenia during Cycles 1-2 | 42-56 days
  Time to recovery of grade 3 neutropenia (absolute neutrophil count<1.0×10^9/L) during Cycles 1-2
Time to recovery of grade 4 neutropenia during Cycles 1-2 | 42-56 days
  Time to recovery of grade 4 neutropenia (absolute neutrophil count <0.5×10^9/L) during Cycles 1-2
Incidence of grade 4 neutropenia during Cycles 1-2 | 42-56 days
  Incidence of grade 4 neutropenia (absolute neutrophil count <0.5×10^9/L) during Cycles 1-2
Incidence of febrile neutropenia during Cycle 2 | 21-28 days
  Incidence of febrile neutropenia during Cycle 2 (i.e., the second chemotherapy cycle post-enrollment)
Proportion of patients with chemotherapy delay or dose reduction in subsequent cycles due to neutropenia during Cycles 1-2 | 42-56 days
  Proportion of patients with chemotherapy delay or dose reduction in subsequent cycles due to neutropenia during Cycles 1-2
Proportion of patients receiving antibiotic treatment and experiencing infections during Cycles 1-2 | 42-56 days
  Proportion of patients receiving antibiotic treatment and experiencing infections during Cycles 1-2

CONTACTS AND LOCATIONS:
Overall Officials: Sidan Li, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No